CLINICAL TRIAL: NCT04547543
Title: Visio-consultation Compared to Face-to-face Consultation During the Follow-up of Apneic Patients Treated by Continuous Positive Airway Pressure (CPAP)
Brief Title: Follow-up of Apneic Patients by Visio-consultation
Acronym: VISIOSAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 38RC19.312
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: Telemedicine; Medical follow-up
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video consultation (Other): Patients in this group will have a continuous positive pressure follow-up visit by videoconsultation
  Interventions: Other: Videoconsultation
- Face-to-face consultation (No Intervention): Patients in this group will have a continuous positive pressure follow-up visit by face-to-face consultation

INTERVENTIONS:
Other: Videoconsultation — Patient randomized on video-consultation group will have a video-consultation with the investigator within 3 months after the randomization. During this consultation, the investigator performs a clinical interrogation in order to collect anthropometric parameters: (sex, age, weight, height, body mass index (BMI)), blood pressure (by blood pressure monitor at home), the level of physical activity (by Actimetry over 7 days), smoking status and alcohol status
  Arms: Video consultation

SUMMARY:
Prospective multicenter open-label randomized clinical trial comparing videoconsultation to a face-to-face consultation during the follow-up of apneic patients treated by continuous positive pressure (CPAP) .

DETAILED DESCRIPTION:
The annual management of Obstructive Sleep Apnea (OSA) patients treated by continuous positive air pressure (CPAP) aims to maintain an optimal level of care while offering to the patients a combined management of their pathology. This management aims to reduce the risk of cardio-metabolic pathologies.

However, the high prevalence of OSA in the general population reduces the ability to explore undiagnosed patients. The contribution of videoconsultation is now available and allows the management of OSA patients treated by CPAP.

The objective of this study is to compare the videoconsultation to a face-to-face consultation during the follow-up of apneic patients treated by continuous positive pressure (CPAP) .

The results of this study could provide very important new data on the impact of videoconsultation on the monitoring a chronic respiratory pathology such as sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* Apneic patient treated with CPAP for more than 12 months and having an annual scheduled follow-up visit.
* Adult patient who can give an informed consent.
* Patient with access to a media (Smartphone, tablet or computer) and an Internet connection at home.

Exclusion Criteria:

* Patient unable to use or understand the digital system.
* Patient under guardianship or deprived of liberty
* Pregnant woman
* Patient in a period of exclusion from another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-09-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Therapeutic adherence to CPAP | 3 months after consultation
  Non inferiority of visioconsultation compared to face-to-face consultation in terms of therapeutic adherence to CPAP evaluated by the difference in compliance 3 months before and 3 months after the consultation
Consultation cost | 3 months after consultation
  Non inferiority of visioconsultation compared to face-to-face consultation in terms of consultation cost evaluated by the difference in cost between the 2 types of consultation
Patient satisfaction: questionnaire | 3 months after consultation
  Non inferiority of visioconsultation compared to face-to-face consultation in terms of patient satisfaction evaluated by the VSQ-VF questionnaire

SECONDARY OUTCOMES:
Sleepiness related to CPAP | 3 and 12 after consultation
  Epworth Sleepiness Scale
Tiredness related to CPAP | 3 and 12 months after consultation
  Pichot's fatigue scale
Evaluate the quality of CPAP treatment (Residual AHI) | 3 and 12 months after consultation
  Evaluate the quality of CPAP treatment by the residual Apnea-Hypopnea Index(AHI) (event/hour)
Evaluate the quality of CPAP treatment (adverse events) | 3 and 12 months after consultation
  Evaluate the quality of CPAP treatment by the adverse event reporting
Evaluate the quality of CPAP treatment (mask leaks level) | 3 and 12 months after consultation
  Evaluate the quality of CPAP treatment by the CPAP mask leaks level (litre/min)
Evaluate the quality of CPAP treatment (visits by the health care provider): number of visits by the health care provider and the reasons for these visits | 3 and 12 months after consultation
  Evaluate the quality of CPAP treatment by collecting the number of visits by the health care provider and the reasons for these visits
Assess the risk factors associated with OSA in patients treated with CPAP (weight) | 12 months after consultation
  Body weight (kg)
Assess the risk factors associated with OSA in patients treated with CPAP (level of physical activity) | 12 months after consultation
  Evaluation of the level of physical activity by actimetry
Assess the risk factors associated with OSA in patients treated with CPAP (blood pressure) | 12 months after consultation
  Blood pressure by blood pressure monitoring at home

CONTACTS AND LOCATIONS:
Overall Officials: Renaud TAMISIER, Pr, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Grenoble-Alpes, Grenoble, France